CLINICAL TRIAL: NCT01575522
Title: A Phase 2 Study of ARQ 197 in Metastatic Triple-negative Breast Cancer
Brief Title: Tivantinib in Treating Patients With Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00722; NCI-2012-00722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DFCI-12-017; CDR0000730102; 12-017 (Other: Dana-Farber Cancer Institute); 8985 (Other: CTEP); P30CA006516 (NIH); U01CA062490 (NIH); NCT01542996 (obsolete NCT alias)
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2015-10

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — ARQ 197

ARMS (1):
- Treatment (tivantinib) (Experimental): Patients receive tivantinib 360 mg PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection at baseline and periodically during study for c-Met expression, relevant markers (HGF and VEGF), PTEN loss, and PI3K mutation analysis by FISH and IHC. Archived tumor tissue samples are also analyzed.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Tivantinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tivantinib — Given PO
  Other Names: ARQ 197; ARQ-197; c-Met Inhibitor ARQ 197

SUMMARY:
This phase II trial studies how well tivantinib works in treating patients with recurrent or metastatic breast cancer. Tivantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the activity of tivantinib (ARQ-197) as defined by 6-month progression-free survival (PFS) of participants with triple-negative metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate objective response based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. To evaluate c-Met and phospho c-Met expression in archival tumor tissue. (Exploratory) III. To evaluate the incidence of c-Met-positive circulating tumor cells at baseline. (Exploratory) IV. To evaluate the effect of ARQ-197 on serum markers relevant to c-Met pathway (hepatocyte growth factor [HGF] and vascular endothelial growth factor [VEGF]). (Exploratory) V. To evaluate phosphatase and tensin homolog (PTEN) loss and PI3K mutations in archival tumor tissue. (Exploratory) VI. To evaluate proportion of participants with basal-like breast cancer. (Exploratory)

OUTLINE: This is a multicenter study.

Patients receive tivantinib orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection at baseline and periodically during study for c-Met expression, relevant markers (HGF and VEGF), PTEN loss, and PI3K mutation analysis by fluorescent in situ hybridization (FISH) and immunohistochemistry (IHC). Archived tumor tissue samples are also analyzed.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with recurrent or metastatic disease; participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Participants must have recent evidence of progressive disease

  * Participants must have received 1-3 prior chemotherapeutic regimens for metastatic breast cancer and must have been off treatment with chemotherapy for at least 14 days before enrollment in the study
* Participants must have discontinued all biologic therapy (including vaccines) at least 14 days before enrollment in the study
* Participants must have discontinued any investigational therapy at least 14 days before enrollment in the study
* Participants may have received prior radiation therapy in either the metastatic or early-stage setting

  * Radiation therapy must be completed at least 14 days before enrollment in the study
  * Participant must not have received radiation to > 25% of his or her bone marrow within 30 days of starting study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 times institutional ULN; for participants with documented liver metastases, AST/ALT =< 5.0 times ULN
* Serum creatinine =< 1.5 times ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Either the primary tumor and/or the metastasis must be triple-negative; the invasive tumor must be hormone-receptor poor, defined as estrogen-receptor negative (ER-) and progesterone-receptor negative (PR-), or staining < 10% by immunohistochemistry (IHC)

  * Human epidermal growth factor receptor 2 (HER2) status: the invasive tumor must be HER2-negative, defined as 0 or 1+ by IHC, or FISH < 2.0
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the study and for 90 days after the last investigational drug dose received
* Female subjects of childbearing potential must have a negative serum pregnancy test within 21 days of cycle 1 day 1
* Participants on bisphosphonates may continue receiving bisphosphonate therapy during study treatment; bisphosphonate therapy may also be initiated on study treatment if needed
* Confirmed availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have received chemotherapy, biologic, investigational, or radiotherapy within 14 days prior to entering the study
* Participants who are receiving any other investigational agents
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms

  * Participants with a history of treated central nervous system (CNS) metastases are eligible

    * Treated brain metastases are defined as those having no evidence of progression or hemorrhage for >= 2 months after treatment, and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging or computed tomography [CT] scan) during the screening period
    * Treatment for brain metastases may include whole-brain radiotherapy, radiosurgery, or a combination as deemed appropriate by the treating physician
  * Participants may be taking anti-convulsant medications, which must be non-enzyme-inducing anti-epileptic drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as >= grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Human immunodeficiency virus (HIV)-positive participants on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute Faulkner Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Tolaney SM, Tan S, Guo H, Barry W, Van Allen E, Wagle N, Brock J, Larrabee K, Paweletz C, Ivanova E, Janne P, Overmoyer B, Wright JJ, Shapiro GI, Winer EP, Krop IE. Phase II study of tivantinib (ARQ 197) in patients with metastatic triple-negative breast cancer. Invest New Drugs. 2015 Oct;33(5):1108-14. doi: 10.1007/s10637-015-0269-8. Epub 2015 Jul 1. PMID 26123926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Tivantinib)
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Tivantinib): Patients receive tivantinib PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection at baseline and periodically during study for c-Met expression, relevant markers (HGF and VEGF), PTEN loss, and PI3K mutation analysis by FISH and IHC. Archived tumor tissue samples are also analyzed.
  Laboratory Biomarker Analysis: Correlative studies
  Tivantinib: Given PO
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20
  Black or African American | 2

OUTCOME MEASURES:

1. Primary Outcome: PFS Status
Description: Analyzed using the Kaplan-Meier method. 95% confidence intervals (CI) will be determined. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from start of treatment to time of progression or death, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 22
months | 1.2 [1.0 to 1.4]

2. Secondary Outcome: Overall Response Using RECIST v1.1
Description: The 95% confidence intervals should be provided. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by Conventional CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >/=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tivantinib)
Number analyzed (Participants) | 22
percentage of participants | 4.5 [0.1 to 22.8]

3. Secondary Outcome: To Evaluate c-Met Expression in Archival Tumor Tissue.
Description: Assessment of ploidy status was done by visual screening of all tumor area; cells with maximum number of signals were recorded. MET amplification was defined as a MET/CEP7 ratio ≥ 2. Samples having a MET/CEP7 ratio from 1.5 and up to 2 were defined as having relative MET gain. Samples with a MET/CEP7 ratio of 1 but with more than two copies of each probe were defined as having polysomy of chromosome 7.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Evaluation of c-Met Positivity: MET amplification was defined as a MET/CEP7 ratio ≥ 2. Samples having a MET/CEP7 ratio from 1.5 and up to 2 were defined as having relative MET gain. Samples with a MET/CEP7 ratio of 1 but with more than two copies of each probe were defined as having polysomy of chromosome 7.
Arm/Group | Evaluation of c-Met Positivity
Number analyzed (Participants) | 22
participants | 10

4. Secondary Outcome: To Evaluate Phospho c-Met Expression in Archival Tumor Tissue.
Description: MET amplification was defined as a MET/CEP7 ratio ≥ 2. Samples having a MET/CEP7 ratio from 1.5 and up to 2 were defined as having relative MET gain. Samples with a MET/CEP7 ratio of 1 but with more than two copies of each probe were defined as having polysomy of chromosome 7.
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Evaluation of Phospho c-Met Positivity: MET amplification was defined as a MET/CEP7 ratio ≥ 2. Samples having a MET/CEP7 ratio from 1.5 and up to 2 were defined as having relative MET gain. Samples with a MET/CEP7 ratio of 1 but with more than two copies of each probe were defined as having polysomy of chromosome 7.
Arm/Group | Evaluation of Phospho c-Met Positivity
Number analyzed (Participants) | 22
participants | 0

5. Secondary Outcome: To Evaluate the Incidence of c-Met Positive Circulating Tumor Cells.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Evaluation of c-Met Positive Circulating Tumor Cells
Number analyzed (Participants) | 7
participants | 1

ADVERSE EVENTS:
Time Frame: April 2012 -
Arm/Group | Treatment (Tivantinib)
Serious Adverse Events (participants affected / at risk) | 13/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivantinib) (N=22)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Neutropenia (Investigations) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Death (General disorders) | 3 (3) — Death due to disease progression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivantinib) (N=22)
Fatigue (General disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less